CLINICAL TRIAL: NCT07238517
Title: Diagnostic Utility of Musculoskeletal Ultrasound in Early Postoperative Evaluation of Posttraumatic Repaired Hand Tendons.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abdelazeem Salah Abdelazeem Rajeh, Principal investigator, Assiut University
Other Study IDs: MSK-US repaired hand tendon
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Ultrasound Evaluation; Hand Tendon Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MSK US — Focus on early postoperative (first 6-12 weeks) assessment after post-traumatic tendon repair.
  Utilization of high-frequency dynamic ultrasound rather than static imaging or delayed MRI.
  Standardized scanning protocol and blinded interpretation to ensure diagnostic validity.
  Designed to evaluate the diagnostic utility of MSK-US compared with conventional clinical follow-up methods.

SUMMARY:
To evaluate the role of musculoskeletal ultrasound in the early postoperative period following hand tendon repair. By assessing its diagnostic accuracy and clinical utility, the study seeks to determine whether routine MSK-US surveillance can contribute to earlier detection of complications, guide timely management decisions, and ultimately improve functional outcomes in patients undergoing hand tendon surgery.

DETAILED DESCRIPTION:
Hand tendon injuries are among the most frequent traumatic lesions of the upper extremity, representing a major cause of emergency and elective surgeries. Despite advances in surgical techniques, these injuries remain challenging due to the risk of postoperative complications such as rupture, adhesions, infection, and impaired tendon gliding. Early recognition of such complications is essential to prevent long-term stiffness, disability, and functional loss .

Postoperative assessment traditionally relies on clinical examination, but this may be limited by pain, swelling, dressings, or poor patient compliance, and subtle complications may not be evident until significant dysfunction develops. Hence, there is a need for a reliable, non-invasive modality to aid early detection and guide timely intervention.

Musculoskeletal ultrasound (MSK-US) has become an important tool for evaluating tendon injuries. It offers high spatial resolution, dynamic real-time imaging, absence of ionizing radiation, cost-effectiveness, and broad availability. In postoperative settings, MSK-US provides valuable information on tendon continuity, vascularity, surrounding soft tissue changes, and the presence of adhesions or fluid collections. Its ability to assess tendon motion dynamically further enhances its role in monitoring functional recovery.

Evidence indicates that MSK-US can detect complications such as rerupture, adhesions, or infection earlier than clinical examination, supporting its role as an adjunctive modality in follow-up. However, standardized use of ultrasound in routine postoperative surveillance of repaired hand tendons has not yet been established.

ELIGIBILITY:
Inclusion Criteria: adults with primary hand tendon repair and able to return for US follow-up.

-

Exclusion Criteria: Patients with collagen disease, congenital hand deformities, bone fractures, revision/staged repairs, active infection/poor wound access, or can't attend follow-up.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who undergone hand tendon repair after trauma
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of musculoskeletal ultrasound (MSK-US) for detecting clinically significant postoperative complications | Up to 12 weeks after surgical repair
  The accuracy of musculoskeletal ultrasound (MSK-US) in identifying clinically significant postoperative complications following surgical repair of posttraumatic hand tendons.
  Complications include rerupture requiring reintervention, deep infection, symptomatic adhesion requiring surgical release, and large seroma or hematoma requiring drainage or evacuation.
  Diagnostic accuracy will be determined by comparing MSK-US findings to a composite clinical reference standard consisting of surgical findings, clinical assessment, and microbiological/imaging confirmation.
  Accuracy measures will include sensitivity, specificity, positive predictive value, negative predictive value, and likelihood ratios.

SECONDARY OUTCOMES:
Time from surgery to detection of postoperative complication by musculoskeletal ultrasound (MSK-US) versus clinical assessment | Up to 12 weeks after surgical repair

CONTACTS AND LOCATIONS:
Overall Officials: Nagham Nabeel Omar, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt